CLINICAL TRIAL: NCT02765165
Title: A Phase 1/2 Dose-escalation of USL311 as Single Agent and in Combination With Lomustine (CCNU) in Subjects With Advanced Solid Tumors, With Subsequent Single Agent and Combination Phase 2 Cohorts for Subjects With Relapsed/Recurrent Glioblastoma Multiforme (GBM)
Brief Title: Phase 1/2 Study of USL311 +/- Lomustine in Advanced Solid Tumors or Relapsed/Recurrent Glioblastoma Multiforme (GBM)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons not related to safety
Sponsor: Proximagen, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P311-201
Record Dates: First submitted 2016-04-19; First posted 2016-05-06 (Estimated); Results first posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Solid Tumors (Phase 1); Relapsed/Recurrent GBM (Phase 2)
Keywords: Phase 1; Phase 2; Glioblastoma Multiforme; Glioblastoma; GBM; Brain Tumor; Brain Cancer; Tumor; Solid Tumor; Tumour; Lomustine; CCNU; CXCR4; Phase 1 Clinical Trial; Phase 2 Clinical Trial
MeSH Terms: conditions — Recurrence; Glioblastoma; Brain Neoplasms; Neoplasms | interventions — Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose-Escalation USL311, Solid Tumor, Part 1a (Experimental): USL311, intravenous, once per week, starting at 60 mg/m˄2
  Interventions: Drug: USL311
- Dose-Escalation USL311, Solid Tumor, Part 1b (Experimental): USL311, oral, daily, starting at 40 mg
  Interventions: Drug: USL311
- Dose-Escalation USL311 with Lomustine, Solid Tumor, Part 2 (Experimental): USL311, oral, daily, starting at dose as determined in Part 1b, in combination with lomustine 90 mg/m˄2, oral, once every 6 weeks
  Interventions: Drug: USL311; Drug: Lomustine
- Dose-Expansion, USL311, GBM, Part 3 (Experimental): USL311, oral, daily, starting at dose determined in Part 1b
  Interventions: Drug: USL311
- Dose-Expansion, USL311 with Lomustine, GBM, Part 4 (Experimental): USL311, oral, daily, in combination with lomustine, oral, once every 6 weeks, at dose(s) as determined in part 2
  Interventions: Drug: USL311; Drug: Lomustine

INTERVENTIONS:
Drug: USL311 — Administered once weekly in a 21-day cycle
  Arms: Dose-Escalation USL311, Solid Tumor, Part 1a
Drug: USL311 — Administered once daily in a 21-day cycle
  Arms: Dose-Escalation USL311, Solid Tumor, Part 1b; Dose-Expansion, USL311, GBM, Part 3
Drug: USL311 — Administered once daily in a 42-day cycle
  Arms: Dose-Escalation USL311 with Lomustine, Solid Tumor, Part 2; Dose-Expansion, USL311 with Lomustine, GBM, Part 4
Drug: Lomustine — Administered once every 6 weeks in a 42-day cycle
  Arms: Dose-Escalation USL311 with Lomustine, Solid Tumor, Part 2; Dose-Expansion, USL311 with Lomustine, GBM, Part 4

SUMMARY:
This is a multicenter, open-label, Phase 1/2, dose-escalation and dose expansion study of a CXCR4 inhibitor, USL311, alone and in combination with lomustine in subjects with advanced solid tumors (Phase 1) and subjects with relapsed/recurrent GBM (Phase 2). The study is designed to explore the safety, tolerability, pharmacokinetics, and preliminary efficacy of USL311 alone and in combination with lomustine.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

1. Provide signed and dated informed consent prior to study-specific screening procedures
2. ≥ 18 years old
3. Karnofsky performance status (KPS) ≥ 70
4. Must have adequate bone marrow and renal/hepatic function within protocol specified limits
5. Disease-free period of > 2 years from any other previous malignancies, excluding curatively treated basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix. Subjects with prostate cancer Stage 1 that do not require treatment may also be included
6. Women and men must use protocol approved methods of contraception
7. Must be able and willing to comply with the study visit schedule and study procedures
8. Must be able to take oral medications
9. Must have available archived tumor tissue and willing and able to provide consent for study access to such tissue
10. For subjects with a history of seizures, must be adequately controlled on a stable regimen of anti-epileptic drugs

    For Phase 1 Subjects Only:
11. Histologically or cytologically documented diagnosis of solid tumor for which no standard therapy is recognized or have failed or intolerant to the standard-of-care treatment
12. Inoperable metastatic or locally advanced, unresectable disease
13. Subjects may have either evaluable or measurable disease
14. Subjects with treated (surgically excised or irradiated) and stable brain metastases are eligible as long as the subject has adequately recovered from treatment and the treatment was ≥ 28 days prior to initiation of study drug(s) and baseline brain computed tomography (CT) with contrast or magnetic resonance imaging (MRI) ≤ 14 days of initiation of study drug is negative for new brain metastases

    For Phase 2 Subjects Only:
15. Histologically confirmed diagnosis of GBM
16. Subjects must have documented recurrence after first-line treatment
17. Prior first-line treatment must have included radiation and temozolomide
18. Subject is suitable for re-resection, per Investigator discretion, as a component of their clinical care
19. No more than one prior resection (Note: biopsy does not count as prior resection)

Exclusion Criteria:

All Subjects

1. Subjects who have had recent systemic anticancer therapies, interventional device treatment and/or radiotherapy either within 14 days prior to first dose of study drug(s) or have not recovered (to grade ≤ 1) from all clinically significant toxicities related to prior therapies
2. Subjects who have had any major surgery (not including re-resection surgery required in Phase 2) within 28 days prior to first dose of study drug(s), or minor surgery within 14 days prior to first day of study drug(s)
3. Subjects taking any strong cytochrome P450 3A4 inducers within 14 days prior to the first dose of study drug(s)
4. Subjects taking any strong cytochrome P450 3A4 inhibitors within 14 days prior to the first dose of study drug(s)
5. Subjects taking any agents with moderate to high risk to prolong QT corrected (QTc) interval or to cause Torsades de Pointes within 14 days prior to the first dose of study drug(s)
6. Subjects who have been treated with an investigational agent or investigational interventional device within 21 days prior to the first dose of study drug(s)
7. Subject is growth factor dependent or transfusion dependent, or has received growth factor support or transfusion support within 14 days prior to the first dose of study drug(s)
8. History of significant cardiac disease
9. Status epilepticus within 1 year prior to the first dose of study drug(s)
10. Pregnant or breastfeeding
11. Any other significant co-morbid conditions that in the opinion of the Investigator would impair study participation or cooperation

    For Phase 1 Subjects Only:
12. Lymphoma as primary cancer

    For Phase 2 Subjects Only:
13. Unable or unwilling to consent to the provision of resected tissue after surgery
14. Prior treatment with plerixafor or another CXCR4 inhibitor
15. Prior treatment with bevacizumab
16. Prior treatment with lomustine and/or carmustine

    For All Cohorts Receiving Oral USL311:
17. Any active medical condition or previous major abdominal surgery or procedure that might, in the investigator's opinion, have a significant effect on USL311 absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tze-Chiang Meng, MD, Study Director — Proximagen, LLC
Locations (6):
- United States (5):
  - Washington University, St Louis, Missouri
  - University of Oklahoma Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Texas/MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - UT Health San Antonio Cancer Center, San Antonio, Texas
- South Texas Accelerated Research Therapeutics (START) - FJD, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled subjects participated in only one part (parts 1, 2, 3 or 4) of the study. Due to early termination of the study, no subjects were enrolled in parts 2, 3 or 4.
Groups:
- Part 1a, Cohort 1: USL311, intravenous, once per week, 60 mg/m˄2, in 21-day cycles
- Part 1a, Cohort 2: USL311, intravenous, once per week, 120 mg/m˄2, in 21-day cycles
- Part 1a, Cohort 3: USL311, intravenous, once per week, 180 mg/m˄2, in 21-day cycles
- Part 1a, Cohort 4: USL311, intravenous, once per week, 250 mg/m˄2, in 21-day cycles
- Part 1b, Cohort 1: USL311, oral, once per day, 40 mg, in 21-day cycles
- Part 1b, Cohort 2: USL311, oral, once per day, 80 mg, in 21-day cycles
- Part 1b, Cohort 3: USL311, oral, once per day, 160 mg, in 21-day cycles
Period: Treatment Period
Arm/Group | Part 1a, Cohort 1 | Part 1a, Cohort 2 | Part 1a, Cohort 3 | Part 1a, Cohort 4 | Part 1b, Cohort 1 | Part 1b, Cohort 2 | Part 1b, Cohort 3
Started | 3 | 4 | 3 | 3 | 6 | 3 | 4
Completed | 0 (Open-ended design for participation until progression or other reason for withdrawal) | 0 (Open-ended design for participation until progression or other reason for withdrawal) | 0 (Open-ended design for participation until progression or other reason for withdrawal) | 0 (Open-ended design for participation until progression or other reason for withdrawal) | 0 (Open-ended design for participation until progression or other reason for withdrawal) | 0 (Open-ended design for participation until progression or other reason for withdrawal) | 0 (Open-ended design for participation until progression or other reason for withdrawal)
Not Completed | 3 | 4 | 3 | 3 | 6 | 3 | 4
Not completed — Progressive disease | 3 | 2 | 3 | 3 | 4 | 2 | 2
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Study terminated | 0 | 0 | 0 | 0 | 0 | 1 | 2
Period: Post-treatment Follow-up
Arm/Group | Part 1a, Cohort 1 | Part 1a, Cohort 2 | Part 1a, Cohort 3 | Part 1a, Cohort 4 | Part 1b, Cohort 1 | Part 1b, Cohort 2 | Part 1b, Cohort 3
Started | 1 (Subjects who chose to enter follow-up, including long term follow-up for survival, after discontinuing treatment. Subjects were not required to enter follow-up.) | 3 (Subjects who chose to enter follow-up, including long term follow-up for survival, after discontinuing treatment. Subjects were not required to enter follow-up.) | 3 (Subjects who chose to enter follow-up, including long term follow-up for survival, after discontinuing treatment. Subjects were not required to enter follow-up.) | 3 (Subjects who chose to enter follow-up, including long term follow-up for survival, after discontinuing treatment. Subjects were not required to enter follow-up.) | 3 (Subjects who chose to enter follow-up, including long term follow-up for survival, after discontinuing treatment. Subjects were not required to enter follow-up.) | 3 (Subjects who chose to enter follow-up, including long term follow-up for survival, after discontinuing treatment. Subjects were not required to enter follow-up.) | 1 (Subjects who chose to enter follow-up, including long term follow-up for survival, after discontinuing treatment. Subjects were not required to enter follow-up.)
Completed | 0 (Open-ended follow-up) | 0 | 0 | 0 | 0 (Open-ended follow-up) | 0 | 0
Not Completed | 1 | 3 | 3 | 3 | 3 | 3 | 1
Not completed — Death | 1 | 2 | 1 | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Site terminated by sponsor | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Initiation of subsequent treatment | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by the sponsor | 0 | 0 | 0 | 0 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 1a, Cohort 3,: USL311, intravenous, once per week, 180 mg/m˄2, in 21-day cycles
- Part 1a, Cohort 4,: USL311, intravenous, once per week, 250 mg/m˄2, in 21-day cycles
- Part 1b, Cohort 1: USL311, oral, daily, 40 mg, in 21-day cycles
- Part 1b, Cohort 2: USL311, oral, daily, 80 mg, in 21-day cycles
- Part 1b, Cohort 3: USL311, oral, daily, 160 mg, in 21-day cycles
- Total: Total of all reporting groups
Arm/Group | Part 1a, Cohort 1 | Part 1a, Cohort 2 | Part 1a, Cohort 3, | Part 1a, Cohort 4, | Part 1b, Cohort 1 | Part 1b, Cohort 2 | Part 1b, Cohort 3 | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 6 | 3 | 4 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 2 | 3 | 1 | 3 | 17
  >=65 years | 0 | 1 | 1 | 1 | 3 | 2 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (24.83) | 53.5 (16.20) | 57.7 (17.79) | 60.3 (10.97) | 62.5 (14.60) | 72.0 (9.17) | 57.3 (6.95) | 58.8 (14.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3 | 3 | 2 | 1 | 12
  Male | 2 | 2 | 3 | 0 | 3 | 1 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 4
  Not Hispanic or Latino | 3 | 3 | 3 | 2 | 5 | 2 | 4 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 3 | 4 | 2 | 2 | 6 | 3 | 3 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 2 | 3 | 6 | 3 | 4 | 25
  Spain | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Body surface area [Mean (Standard Deviation); unit: m^2] | 1.767 (0.0503) | 2.018 (0.3363) | 2.000 (0.2307) | 1.787 (0.1704) | 1.910 (0.3864) | 1.820 (0.0624) | 2.088 (0.1893) | 1.923 (0.2603)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the highest safe dose (mg/m^2) administered where safe is defined by having at least a 50% probability that the dose limiting toxicity (DLT) rate is less than 33%, as determined by a modified continuous reassessment model.
Time Frame: Assessed weekly during treatment period. Median duration of exposure was 5.14 (range 2.1-17.3) weeks.
Measure: Number; unit: mg/m^2
Groups:
- Part 1a, Dose-escalation, All Oral Cohorts: USL311, intravenous, once per week, starting at 60 mg/m˄2, in 21-day cycles
Arm/Group | Part 1a, Dose-escalation, All Oral Cohorts
Number analyzed (Participants) | 13
mg/m^2 | NA — An MTD was not determined for Part 1a due to early termination of intravenous dosing and change to oral dosing

2. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the highest safe dose (mg) administered where safe is defined by having at least a 50% probability that the dose limiting toxicity (DLT) rate is less than 33%, as determined by a modified continuous reassessment model.
Time Frame: Assessed weekly during treatment period. Median duration of exposure was 6.00 (range 0.3-30.0) weeks.
Measure: Number; unit: mg
Groups:
- Part 1b, Dose-escalation, All Oral Cohorts: USL311, oral, once per day, starting at 40 mg, in 21 day cycles
Arm/Group | Part 1b, Dose-escalation, All Oral Cohorts
Number analyzed (Participants) | 13
mg | NA — An MTD was not determined in Part 1b due to study termination

3. Secondary Outcome: Percentage Progression Free Survival (PFS) at 6 Months (PFS-6m)
Description: Percentage of subjects who were without progression at 6 months as assessed radiographically with response to treatment determined by Response Evaluation Criteria in Solid Tumors (RECIST) or Response Assessment in Neuro-Oncology (RANO) criteria.
Time Frame: Once every 6 weeks during treatment
Population: Due to early termination of study in Phase 1, efficacy outcomes, including PFS-6m, were not analyzed for subjects in Part 1a or Part 1b. Therefore no subjects were included in this analysis population.
Groups:
- Part 1, Dose-escalation, All Cohorts: USL311, intravenous once per week, starting at 60 mg/m˄2, or oral once per day, starting at 40 mg, in 21-day cycles
Arm/Group | Part 1, Dose-escalation, All Cohorts
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Percentage of subjects alive five years after start of treatment.
Time Frame: Weekly during treatment or every 12 weeks during follow-up
Population: Due to early termination of study in Phase 1, efficacy outcomes, including OS, were not analyzed for subjects in Part 1a or Part 1b. Therefore no subjects were included in this analysis population.
Arm/Group | Part 1, Dose-escalation, All Cohorts
Number analyzed (Participants) | 0

5. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Time after initiation of treatment before disease progression
Time Frame: Every 6 weeks during treatment
Population: Due to early termination of study in Phase 1, efficacy outcomes, including median PFS, were not analyzed for subjects in Part 1a or Part 1b. Therefore no subjects were included in this analysis population.
Arm/Group | Part 1, Dose-escalation, All Cohorts
Number analyzed (Participants) | 0

6. Secondary Outcome: Objective Response Rate (ORR%)
Description: Percentage of patients whose disease decreased (Partial response) and/or disappears (Complete response) after initiation of treatment
Time Frame: Every 6 weeks
Population: Number of participants changed to 0 and explanation modified to "Due to early termination of study in Phase 1, efficacy outcomes, including ORR% were not analyzed for subjects in Part 1a or Part 1b. Therefore no subjects were included in this analysis population.
Arm/Group | Part 1, Dose-escalation, All Cohorts
Number analyzed (Participants) | 0

7. Secondary Outcome: Peak Concentration (Cmax)
Description: Peak USL311 concentration (Cmax) in plasma
Time Frame: Day 1
Population: Subjects who received scheduled dose and had sufficient PK samples for determination of parameters
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 1a, Cohort 1: USL311, intravenous, once per week over 2 hours, 60 mg/m˄2, in 21-day cycles
- Part 1a, Cohort 2: USL311, intravenous, once per week over 2 hours, 120 mg/m˄2, in 21-day cycles
- Part 1a, Cohort 3a: USL311, intravenous, once per week over 2 hours, 180 mg/m˄2, in 21-day cycles
- Part 1a, Cohort 3b: USL311, intravenous, once per week over 4 hours, 180 mg/m˄2, in 21-day cycles
- Part 1a, Cohort 4: USL311, intravenous, once per week over 4 hours, 250 mg/m˄2, in 21-day cycles
Arm/Group | Part 1a, Cohort 1 | Part 1a, Cohort 2 | Part 1a, Cohort 3a | Part 1a, Cohort 3b | Part 1a, Cohort 4 | Part 1b, Cohort 1 | Part 1b, Cohort 2 | Part 1b, Cohort 3
Number analyzed (Participants) | 3 | 4 | 1 | 2 | 2 | 5 | 3 | 4
ng/mL | 48.2 (41.1) | 69.1 (66.9) | 200 (NA) — CV% not calculable as 1 subject | 168 (94) | 107 (37.2) | 2.06 (84.6) | 4.74 (32.4) | 6.68 (58.5)

8. Secondary Outcome: Time to Peak Concentration (Tmax)
Description: Time to peak concentration of USL311 in plasma
Time Frame: Day 1
Population: Subjects who received scheduled dose and had sufficient PK samples for determination of parameters
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1a, Cohort 1 | Part 1a, Cohort 2 | Part 1a, Cohort 3a | Part 1a, Cohort 3b | Part 1a, Cohort 4 | Part 1b, Cohort 1 | Part 1b, Cohort 2 | Part 1b, Cohort 3
Number analyzed (Participants) | 3 | 4 | 1 | 2 | 2 | 5 | 3 | 4
Hours | 1.05 [1.02 to 2.03] | 1.04 [1.02 to 2.03] | 0.53 [0.53 to 0.53] | 2.28 [0.5 to 4.05] | 2.55 [2.05 to 3.05] | 0.63 [0.48 to 2] | 0.67 [0.53 to 1] | 0.565 [0.52 to 0.98]

9. Secondary Outcome: Area Under the Concentration Versus Time Curve (AUC)
Description: Area under the curve versus time from time 0 to infinity for USL311 concentration in plasma
Time Frame: Day 1
Population: Subjects who received scheduled dose and had sufficient PK samples for determination of parameters
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part 1a, Cohort 1 | Part 1a, Cohort 2 | Part 1a, Cohort 3a | Part 1a, Cohort 3b | Part 1a, Cohort 4 | Part 1b, Cohort 1 | Part 1b, Cohort 2 | Part 1b, Cohort 3
Number analyzed (Participants) | 3 | 4 | 1 | 2 | 2 | 5 | 3 | 4
ng*h/mL | 181 (101) | 437 (16.7) | 711 (NA) — CV% not calculable as 1 subject | 1193 (48.3) | 1059 (15.3) | 5.95 (54.1) | 16.4 (51) | 30.4 (56.3)

ADVERSE EVENTS:
Time Frame: Adverse events collected from informed consent to last visit during treatment period (post treatment follow-up visit or end of treatment visit, whichever was last). Median duration of exposure was 5.14 (range 2.1-17.3) weeks for Part 1a (intravenous) subjects and 6.00 (range 0.3-30.0) for Part 1b (oral) subjects. Survival information only was collected during long term follow-up; for those who entered follow-up, follow-up was up to 25 months in Part 1a and up to 16 months in Part 1b.
Description: Study visits once per week during Treatment with adverse event collection, vital sign measurements, physical examination, neurologic examination and laboratory assessments at each visit. Safety electrocardiograms once per week first two 21-day cycles and then at beginning of each cycle and at the End of Treatment Visit. Survival information only was collected quarterly during long term follow-up. Deaths during follow-up phase were not captured as serious adverse events unless considered related.
Groups:
- Part 1a, Cohort 1: USL311, intravenous, once per week, at 60 mg/m˄2, in 21-day cycles
- Part 1a, Cohort 2: USL311, intravenous, once per week, at 120 mg/m˄2, in 21-day cycles
- Part 1a, Cohort 3: USL311, intravenous, once per week, at 180 mg/m˄2, in 21-day cycles
- Part 1a, Cohort 4: USL311, intravenous, once per week, at 250 mg/m˄2, in 21-day cycles
Arm/Group | Part 1a, Cohort 1 | Part 1a, Cohort 2 | Part 1a, Cohort 3 | Part 1a, Cohort 4 | Part 1b, Cohort 1 | Part 1b, Cohort 2 | Part 1b, Cohort 3
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/4 | 1/3 | 1/3 | 1/6 | 1/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/4 | 0/3 | 1/3 | 3/6 | 1/3 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/4 | 1/3 | 3/3 | 6/6 | 3/3 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1a, Cohort 1 (N=3) | Part 1a, Cohort 2 (N=4) | Part 1a, Cohort 3 (N=3) | Part 1a, Cohort 4 (N=3) | Part 1b, Cohort 1 (N=6) | Part 1b, Cohort 2 (N=3) | Part 1b, Cohort 3 (N=4)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1a, Cohort 1 (N=3) | Part 1a, Cohort 2 (N=4) | Part 1a, Cohort 3 (N=3) | Part 1a, Cohort 4 (N=3) | Part 1b, Cohort 1 (N=6) | Part 1b, Cohort 2 (N=3) | Part 1b, Cohort 3 (N=4)
Electrocardiogram QT prolonged (Investigations) | 0 | 2 | 1 | 2 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorders (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Cervical cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Small cohort sample size. Heterogenous solid tumor types.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to first publication which is intended to be a joint, multi-center publication in conjunction with the Investigators. Following first publication, the Investigator may publish results provided the proposed publication is submitted for review to the Sponsor at least 60 days in advance; the Sponsor has the right to remove confidential/proprietary information. If publication may affect patentability of an invention, an additional delay of 90 days may be requested.

DOCUMENTS (2):
  • Study Protocol (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT02765165/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT02765165/SAP_001.pdf